CLINICAL TRIAL: NCT06616428
Title: Acute Effects of Commercial Group Exercise Classes on Arterial Stiffness and Cardiovagal Modulation in Healthy Young and Middle-aged Adults: an Ecological Valid Model
Brief Title: Acute Exercise Effects on Arterial Stiffness and Cardiovagal Modulation in Adults
Acronym: PUMPING ARTERY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egas Moniz - Cooperativa de Ensino Superior, CRL (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: PUMPING ARTERIES
Record Dates: First submitted 2024-09-22; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Ageing; Aerobic Exercise; Resistance Exercise; Combined Exercise
Keywords: Arterial stiffness; Cardiac autonomic function; Group exercise; Age differences; Ecological validity

STUDY DESIGN:
Intervention Model Description: Parallel group crossover randomized trial
Who Masked: Participant, Care Provider
Masking Description: Outcomes were assed by the same experts in every time point. Participants, evaluators and fitness instructors were blinded until arrival of the participant for each visit.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Aerobic Exercise (Experimental)
  Interventions: Other: Bike group fitness class
- Resistance Exercise (Experimental)
  Interventions: Other: Pump Power
- Combined Exercise (Experimental)
  Interventions: Other: Global Training
- Control (No Intervention)

INTERVENTIONS:
Other: Bike group fitness class — Comprised a rhythmic indoor cycling session, characterized by fluctuations in intensity corresponding to changes in position, music rhythm, cadence, and revolutions per minute. Participants were instructed to strictly follow verbal cues from the instructor, adjusting cycling cadence and resistance as directed, for 45 minutes.
  Arms: Aerobic Exercise
Other: Pump Power — Entails a comprehensive total-body weight-training program with a focus on improving strength, muscular endurance, and overall fitness of large muscle groups. The class, choreographed to music, involved participants performing a combination of barbell, body-weight exercises, and free-weight plates, during 45 minutes. Participants selected weights based on the target muscle group for the specific song or track and their individual fitness goals.
  Arms: Resistance Exercise
Other: Global Training — Incorporated both aerobic and resistance components, combining athletic movements like running, lunging, and jumping with strength exercises such as barbells, body-weight exercises, and free-weight plates for the large muscle groups, during 45 minutes.
  Arms: Combined Exercise

SUMMARY:
Background and Gap:

The physiological importance of large artery distensibility in cardiovascular function is well-established. Stiffening of central arteries leads to elevated systolic blood pressure (SBP), increased left ventricular afterload, and altered coronary artery perfusion. These changes can elevate cardiovascular disease risk and all-cause mortality. Cardiac autonomic function, including heart rate recovery (HRR) and heart rate variability (HRV), is closely linked to blood pressure regulation. Reductions in HRR and HRV are predictive of cardiovascular mortality. The dynamic regulation of arterial stiffness and autonomic function post-exercise is crucial for both health and performance outcomes. Exercise, particularly aerobic, has been shown to reduce arterial stiffness, but evidence across different exercise modalities is limited, especially for group fitness classes. These classes are a common method for achieving cardiovascular fitness, but their acute effects on arterial stiffness and autonomic function remain understudied.

Study Type: Parallel Group Crossover Randomised Trial Primary Purpose: To assess and compare the acute effects of three commercially available group exercise classes on arterial stiffness and cardiovagal modulation in healthy young and middle-aged adults.

Study Population: Healthy adults aged 18-60 years.

Main Question:

How does age influence post-exercise recovery patterns in arterial stiffness and cardiovagal modulation following different group fitness classes?

Comparison Group: Researchers compared arterial stiffness and autonomic function responses across three group fitness classes in young and older adults.

Participant Tasks:

* Attend a 60-minute group exercise class.
* Undergo measurements of arterial stiffness and autonomic function before and after 3 group fitness classes.

DETAILED DESCRIPTION:
All participants were randomly assigned to 1 of 4 experimental conditions using a randomized block scheme (https://www.randomizer.org/). Participants completed 4 separate intervention sessions, each consisting of an initial rest, a group fitness class of either indoor cycling, resistance training, combined exercise training, or no exercise (CON), followed by a recovery period. A minimum of 72 hours between sessions was ensured. Body composition and cardiorespiratory fitness for each participant were evaluated before and after the CON session, respectively.

Each session began with 20 minutes of supine rest on a cushioned examination table, with resting energy expenditure (REE) measured by indirect calorimetry (K5, Cosmed, Rome, Italy) and heart rate (HR) and blood pressure (BP) recorded continuously using digital plethysmography (Finapres, NOVA, Finapres Medical Systems, Amsterdam, The Netherlands). This was followed by: 1) Regional assessments of PWV and pulse wave analysis of the carotid, brachial, femoral, and distal arteries on the right side of the body using applanation tonometry (Complior 2.0, Alam Medical; Saint Quentin Fallavier, France); and 2) Assessment of heart rate variability (HRV) and baroreflex sensitivity (BRS) indices using the Finapres NOVA 5 ECG lead module. Following these assessments, participants engaged in a 45-minute group fitness class, while activity energy expenditure (AEE) was continuously measured by indirect calorimetry (K5, Cosmed, Rome, Italy). In the CON session, participants remained comfortably seated for 45 minutes, maintaining a good posture. After each group fitness class, participants immediately returned to the examination table and recovered in the supine position for 30 minutes, during which local and regional stiffness, HRV, and baroreflex sensitivity (BRS) were re-evaluated at 10-, 20-, and 30-minute intervals during recovery and compared to those at rest. Participants were blinded to the order of the experimental interventions until arrival at the laboratory. All sessions were conducted in the morning to minimize potential diurnal variation. Participants were also instructed not to ingest any food or drink (except water) 4 hours before the sessions and to avoid alcohol, caffeine, and exercise for at least 24 hours preceding each session.

Based on a medium effect size of 0.154 derived from published changes in aortic PWV within-between modes of exercise (23), an a priori power analysis suggested that 22 participants were required (11 per group) to detect significant differences within-between groups, conditions, and time points (1-β = 80%, α = 0.05).

ELIGIBILITY:
Inclusion Criteria:

* Physically active, as assessed by the International Physical Activity Questionnaire (IPAQ)
* Experience in both aerobic and resistance exercise (∼3-4 times/week, for more than 3 months).
* Healthy or perceived to be healthy based on the sport's medical examination or the preparticipation screening process, Physical Activity Readiness Questionnaire for Everyone (PARQ+).

Exclusion Criteria:

* Any form of cardiovascular disease
* More than one cardiovascular disease risk factor
* Resting hypertension (SBP >140 mmHg, DBP > 90 mmHg)
* Any prescription medication use that may influence vascular and autonomic response to exercise
* Being an athlete
* Currently smoking.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2021-11-26 (Actual); Study Completion 2022-03-11 (Actual)

PRIMARY OUTCOMES:
Changes in Blood Pressure | Evaluations were conducted at rest before exercise, and at 10, 20, and 30 minutes post-exercise
  Resting brachial blood pressures (systolic and diastolic) were measured in the supine position using an automated oscillometric cuff (HEM-907 XL; Omron Corporation, Japan). Two measurements were taken, and the average was recorded for analysis. Pulse pressure was calculated as the difference between systolic and diastolic blood pressure. Central blood pressure was assessed by applanation tonometry (Complior 2.0, Alam Medical; Saint Quentin Fallavier, France) from right carotid traces obtained during carotid-femoral pulse wave velocity assessment. The waveforms were averaged, and mean values were taken from a 15-second acquisition window. Carotid waveforms were calibrated using mean arterial pressure measured just before acquisition.
Changes in Heart Rate Variability | Evaluations were conducted at rest before exercise, and at 10, 20, and 30 minutes post-exercise
  R-R intervals were sampled at 300 Hz using a 5-ECG lead module (Finapres Nova, Finapres Medical Systems). Heart rate variability analyses were conducted offline with FisioSinal software in Matlab. After detecting R-R peaks and removing artifacts, 2-minute time series were created using cubic spline interpolation to estimate time-domain and spectral power indices. Ectopic heartbeats (mean = 1, SD = 6 bpm) were excluded. Time-domain indices included SDNN (overall variability) and RMSSD (cardiovagal modulation). Daubechy-12 wavelet analysis estimated low-frequency (vagal/sympathetic) and high-frequency (cardiovagal) bands.
Changes in Cardiovagal Baroreflex Sensitivity | Evaluations were conducted at rest before exercise, and at 10, 20, and 30 minutes post-exercise
  Baroreceptor Sensitivity was estimated using the spontaneous sequence method in FisioSinal, focusing on SBP (more than 1 mmHg) and RR interval (more than 4 ms) ramps. SBP was recorded using finger plethysmography (Finapres® NOVA).
Changes in Regional Arterial Stiffness | Evaluations were conducted at rest before exercise, and at 10, 20, and 30 minutes post-exercise
  Pressure waveforms from the carotid, femoral, radial, and distal arteries were captured simultaneously using applanation tonometry (Complior 2.0, Alam Medical; Saint Quentin Fallavier, France). The distance between pulse sites was measured and entered into the software, with carotid-femoral distance corrected by a 0.8 factor. Sensors were positioned for the carotid and radial arteries, while femoral and distal posterior tibial arteries were held manually. After obtaining 10 carotid pulse waveforms, simultaneous recording of carotid, femoral, radial, and distal posterior tibial pressure curves occurred. Transit time between waveforms was calculated using the foot-to-foot algorithm. Pulse wave velocity from carotid to femoral, carotid to radial, and carotid to distal posterior tibial arteries were used as indices of central and peripheral arterial stiffness.

SECONDARY OUTCOMES:
Energy Expenditure | Before and throughout the group fitness classes
  For the resting energy expenditure (REE) assessment, participants arrived 60 minutes before each session after a 2-3 hour fast. After 10 minutes of seated rest in a dimly lit room, REE was measured for 15 minutes using indirect calorimetry (K5, Cosmed, Rome, Italy). VO2, CO2, respiratory exchange ratio, and ventilation were continuously collected and averaged over 1-minute intervals. The first 5 minutes of data were discarded, and the mean of a 5-minute steady-state interval, where RER ranged from 0.7 to 1.0, was used to calculate REE. The mean VO2 and CO2 during this steady state were applied to the Weir equation, and the lowest REE period was used.
  VO2 was also measured throughout the session for total energy expenditure (TEE) analysis. Activity energy expenditure (AEE) was calculated as TEE minus REE and 0.1*TEE. REE was also used to calculate intensities in metabolic equivalents.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Melo, PhD, Principal Investigator — Egas Moniz School of Health & Science
Locations (1):
- Ginásio Clube Português, Lisbon, Lisbon District, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Data obtained in this study may be provided to qualified researchers with academic interest in vascular responses to resistance training with blood flow restriction. Data or samples shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol
Time Frame: Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact xmelo@egasmoniz.edu.pt

REFERENCES:
- [Background] Maroco JL, Pinto M, Laranjo S, Santa-Clara H, Fernhall B, Melo X. Cardiovagal Modulation in Young and Older Male Adults Following Acute Aerobic Exercise. Int J Sports Med. 2022 Oct;43(11):931-940. doi: 10.1055/a-1843-7974. Epub 2022 May 4. PMID 35508200
- [Background] Cunha FA, Midgley AW, Goncalves T, Soares PP, Farinatti P. Parasympathetic reactivation after maximal CPET depends on exercise modality and resting vagal activity in healthy men. Springerplus. 2015 Feb 27;4:100. doi: 10.1186/s40064-015-0882-1. eCollection 2015. PMID 25793148
- [Background] Ashor AW, Lara J, Siervo M, Celis-Morales C, Mathers JC. Effects of exercise modalities on arterial stiffness and wave reflection: a systematic review and meta-analysis of randomized controlled trials. PLoS One. 2014 Oct 15;9(10):e110034. doi: 10.1371/journal.pone.0110034. eCollection 2014. PMID 25333969
- [Background] Michael S, Graham KS, Davis GM Oam. Cardiac Autonomic Responses during Exercise and Post-exercise Recovery Using Heart Rate Variability and Systolic Time Intervals-A Review. Front Physiol. 2017 May 29;8:301. doi: 10.3389/fphys.2017.00301. eCollection 2017. PMID 28611675
- [Derived] Melo X, Lopes A, Coelho R, Simao B, Oliveira I, Maroco JL, Laranjo S, Fernhall B, Santa-Clara H. Acute effects of commercial group exercise classes on arterial stiffness and cardiovagal modulation in healthy young and middle-aged adults: A crossover randomized trial. PLoS One. 2025 Mar 13;20(3):e0319130. doi: 10.1371/journal.pone.0319130. eCollection 2025. PMID 40080484